CLINICAL TRIAL: NCT02444910
Title: Effects of KDT501 on Metabolic Features in Insulin Resistant Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: KinDex Pharmaceuticals, Inc. (Industry)
Collaborators: University of Kentucky (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8265426; Product IND Number: 113,652 (Other: FDA)
Record Dates: First submitted 2015-05-07; First posted 2015-05-15 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: KDT501; Diabetes; Diabetes Mellitus; Type 2; KinDex
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- KDT501 (Experimental): Experimental drug, KDT501, is administered at 600mg for 10 consecutive days. On days 11 and 21 (+/- 1 day), based on the KDT501 drug exposure level, the subject will be provided instructions on dose adjustment of KDT501. Dose adjustments will be administered at 800mg for 10 consecutive days, determined at day 11; followed by 1,000mg for 8 consecutive days if determined at day 21.
  Interventions: Drug: KDT501

INTERVENTIONS:
Drug: KDT501 — 600mg twice daily, Oral, for 10days; then 800mg twice daily, Oral, for 10 days; then 1,000mg twice daily, Oral, for 8 days.

SUMMARY:
KDT501 is an orally administered product designed to help control impaired glucose and insulin regulation in patients with insulin resistance. Nonclinical studies demonstrate agonist activity of KDT501 at the G-protein coupled receptor 120 as well as other G-protein receptors. Nonclinical studies have also documented the ability of KDT501 to improve insulin sensitivity and glucose regulation as well as reduce proinflammatory signals. These properties combined with antihyperglycemic activity and modest, partial agonist effect of KDT501 at the peroxisome proliferator-activated receptor-gamma (PPARγ) receptor suggests an atypical and pleiotropic mechanism of action for KDT501.

Following providing informed consent, potential subjects will undergo screening procedures to ensure that they meet all inclusion and exclusion criteria. Following registration on study, subjects will undergo baseline pretreatment studies, including two abdominal fat biopsies, one taken after cold challenge, as well as determination of resting metabolic rate, a 4 hour lipid tolerance test, and a 2 hour euglycemic clamp study. All pretreatment studies in registered subjects will be performed within 7 days prior to initiating therapy. On the first day of treatment (Day 0), subjects will take the first 600 mg dose of KDT501 in the clinic, followed by serum pharmacokinetic (PK) samples being obtained every hour for 6 hours after dosing. Subjects will then continue dosing as an outpatient, 600 mg po twice daily. All doses will be taken with meals (breakfast and dinner). On Day 7, subjects will return to the clinic to undergo safety and laboratory assessments, including PK. On Days 14 and 21, subjects will again return to the clinic to undergo safety and laboratory assessments. On Day 17 subjects will return to the clinic for PK studies, as noted below. Treatment in all subjects will end on Day 28. Rapid PK assessment of drug exposure, defined as AUC0-12h, will be performed following PK samples drawn at Time 0, 1h, 2h, 3h, 4h, 5h, 6h, 8h, 10h, and 12h on both Days 7 and 17. On Days 11 and 21 (±1day), based on the KDT501 drug exposure level, the subject will be provided instructions on dose adjustments of KDT501. The maximum allowed KDT501 exposure ceiling for all subjects enrolled is AUC0-12h = 22,500ng-hr/mL.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained prior to the initiation of study procedures
2. Age is 40-70 years
3. Diagnosis IGT, IFG, or metabolic syndrome

   * IGT is defined as: a) 2 hour OGTT glucose 140-199mg/dL and b) fasting glucose <126 mg/dL
   * IFG is defined as: a) 2 hour OGTT glucose < 200 mg/dL and b) fasting glucose 100-125 mg/dL
   * Metabolic syndrome is defined as meeting at least 3 of the following criteria: a) serum triglycerides >150 mg/dL; b) serum HDL<40 mg/dl (males) or <50 (females); c) BP>130/85 or on medical treatment; d) waist circumference >40" (males) or >35" (females); e)HbA1c>5.7%
4. Prior therapy for IGT and IFG may include diet alone
5. HbA1c <7.0% within 28 days of registration
6. Fasting plasma glucose <126 mg/dL within 28 days of registration
7. Body mass index (BMI) ≥27 kg/m2
8. Women of child-bearing potential have a negative serum pregnancy test result ≤28 days prior to registration and agree not to breastfeed during investigational treatment with KDT501 and for 28 days following the final dose of KDT501.
9. All males and premenopausal females who have not been surgically sterilized have agreed to practice a method of birth control considered by the Investigator to be effective and medically acceptable for at least 14 days prior to registration, throughout treatment, and for 28 days following the final dose of KDT501.
10. Adequate baseline hematologic, renal, and liver function as evidenced by laboratory test results within the following ranges (obtained ≤28 days prior to registration):

    * Hemoglobin >11.0 gm/dL
    * Platelet Count ≥100 x 10^3/μL
    * White Blood Count ≥2.0 x 103/μL and ≤15.0 x 103/μL
    * Creatinine Clearance ≥60 mL/min
    * Total Bilirubin ≤2 x upper limit of normal (ULN)
    * Aspartate Transferase (AST) ≤2.5 x ULN
    * Alanine Transferase (ALT) ≤2.5 x ULN
    * INR< 1.5 and PTT <1.5 ULN
11. World Health Organization (WHO) performance status 0-1

Exclusion Criteria:

1. Prior or current history of T2DM
2. Type 1 diabetes
3. Subjects with IGT or IFG who have hypoglycemic unawareness and/or recurrent severe hypoglycemia
4. NYHA CHF Class 2-4
5. Any significant, active pulmonary disorder including FEV1 <60% predicted based on outpatient spirometry
6. History of any significant cardiovascular disease, including arrhythmia, clinically significant ECG abnormality, uncontrolled hypertension, myocardial infarction or unstable angina pectoris within the past 6 months
7. History of HIV or AIDS
8. Active Hepatitis B or C infection requiring therapy within the past 6 months
9. History of any significant, active gastrointestinal disorder, including GERD>grade 2 severity
10. History of gastrectomy or any other GI tract surgery that may affect digestion or absorption
11. Positive fecal occult blood
12. Concomitant therapy with anticoagulants, aspirin or aspirin containing products. Low dose aspirin (≤81 mg qd) is allowed if PT/INR and aPTT values are WNL.
13. Any significant, active hematological disorder
14. Concomitant therapy with CYP2C9 substrates or inhibitors
15. Any major surgery (e.g., surgery requiring general anesthesia) ≤28 days prior to registration
16. Systemic treatment on any investigational clinical trial ≤28 days prior to registration
17. Systemic glucocorticoid or immunosuppressive therapy use ≤28 days prior to registration. Use of a short course (i.e., ≤1 day) of a glucocorticoid is acceptable to prevent a reaction to IV contrast used for CT scans. Topical and inhaled steroid medications are allowed.
18. Any infection requiring parenteral antibiotic therapy or causing fever (i.e., temperature >100.5°F or >38.1°C) ≤7 days prior to registration
19. A contraindication to the use of KDT501
20. Any medical intervention, has any other condition, or has any other circumstance which, in the opinion of the Investigator or the KinDex Medical Monitor, could compromise adherence with study requirements or otherwise compromise the study's objectives

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-04; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline of the 2 hour oral glucose tolerance test (OGTT) at day 28. | 28 days (± 2 days)
  The change in serum glucose 2 hours following the administration of 75gm of oral glucose (2 hour oral glucose tolerance test (OGTT)) will be calculated as the difference in 2 hour OGTT at Day 28 (±2 days) vs. baseline.

SECONDARY OUTCOMES:
Change in Resting Metabolic Rate (RMR) | 27 days (±4 days)
  The change in RMR will be calculated as the difference in RMR at Day 27 (±4 days) vs. baseline.
Change in Lipid Tolerance Test | 27 days (±4 days)
  The change in lipid tolerance test parameters will be calculated as the difference at Day 27 (±4 days) vs. baseline.
Change in HbA1c, fructosamine, and glycated albumin | 27 days (±4 days)
  The change in each of these assay results will be calculated as the difference at Day 27 (±4 days) vs. baseline.
Change in Fasting Plasma Glucose | 27 days (±4 days)
  The change in fasting plasma glucose will be calculated as the difference at Day 27 (±4 days) vs. baseline.
Change in Insulin Sensitivity Based on Euglycemic Clamp Study | 27 days (±4 days)
  The change in insulin sensitivity will be calculated as the difference at Day 27 (±4 days) vs. baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Kern, MD, Principal Investigator — University of Kentucky's Center for Clinical and Translational Science (CCTS)
Locations (1):
- University of Kentucky's Center for Clinical and Translational Science (CCTS), Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Finlin BS, Zhu B, Kok BP, Godio C, Westgate PM, Grayson N, Sims R, Bland JS, Saez E, Kern PA. The Influence of a KDT501, a Novel Isohumulone, on Adipocyte Function in Humans. Front Endocrinol (Lausanne). 2017 Sep 29;8:255. doi: 10.3389/fendo.2017.00255. eCollection 2017. PMID 29033896